CLINICAL TRIAL: NCT02663934
Title: Exercise Training to Improve Brain Health in Older HIV+ Individuals
Acronym: Ex/HIV
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 Risk
Sponsor: Washington University School of Medicine (Other)
Collaborators: University of Missouri, St. Louis (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 201508002
Record Dates: First submitted 2016-01-09; First posted 2016-01-26 (Estimated); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-02

CONDITIONS: HIV
Keywords: HIV, AIDS, Cognition, Memory, Exercise, Stretching
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Motor Activity | interventions — Exercise; Drug Interactions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Exercise (EXS) (Experimental): All EXS sessions will be at an exercise facility at the WUSTL medical campus. Sessions will be offered weekdays. Each session will start with range of motion exercises. Participants will follow an individualized exercise training prescription based on baseline cardiovascular testing. Individual aerobic exercise intensity is based on % of maximum heart rate achieved during the baseline cardiorespiratory fitness test. The target exercise HR will start at 50% and progress to 85% HR reserve. During aerobic exercise, a battery-operated HR monitor will monitor HR. Exercise intensity & duration will be increased as the participant acclimates to the exercise prescription. Adaptation is determined when a given exercise intensity yields a lower HR than prior sessions conducted at the same intensity.
  Interventions: Behavioral: Exercise
- Social Interaction Stretching (SIS) (Active Comparator): This group will serve as a control group against which to gauge the effects of aerobic and resistance training on cognitive function. Participants in this group will follow the same schedule and format as the EXS group. These participants will be supervised by the same trainer and will receive the same amount of attention and class interaction as participants in the EXS program. These SIS participants will receive instructions on stretching, range of motion, limbering, and toning; but the intensity will be far less than that achieved in the EXS classes. Activities will focus on flexibility enhancement. As the participant's level of flexibility increases, stretches with increasing levels of difficulty will be incorporated into the program.
  Interventions: Behavioral: Stretching and Social Interaction

INTERVENTIONS:
Behavioral: Exercise — The resistance exercise training component will follow aerobic exercise and will consist of 4 upper and 3 lower body routines. A combination of guided-motion machines and free weights will be used. Voluntary maximum strength will be measured during the first 4 sessions on each exercise station. The program will initially consist of 1-2 sets of each exercise while lifting a weight that causes muscle fatigue after 8-10 repetitions. The trainer will monitor each participant's exercise response, and when the participant can comfortably lift the weight for 12 repetitions on any exercise, the weight will be increased to cause the muscle group to fatigue after 8 repetitions. This progressive 8-12 repetition cycle is repeated for each exercise over 26 weeks.
  Arms: Exercise (EXS)
Behavioral: Stretching and Social Interaction — Participants will receive instructions on stretching, range of motion, limbering, and toning. Activities will focus on flexibility enhancement. Along with the stretching and flexibility, this group will have a social interaction component. They will have discussions and interact with trainers and coordinators during all their sessions. These participants will be supervised by the same trainer and will receive the same amount of attention and class interaction as participants in the EXS program.
  Arms: Social Interaction Stretching (SIS)

SUMMARY:
Management and treatment of older persons living with HIV (PLWH) (≥ 40 years old) is becoming increasingly more complex as a majority is greater than 40 years old. This proposal will conduct a prospective controlled intervention trial to assess the quantitative and qualitative effects of a monitored aerobic/resistance exercise (EXS) program compared to a social-interaction stretching (SIS) program on brain health (neuropsychological performance testing and neuroimaging measurements) in older PLWH. These results could influence public health policy by encouraging PLWH to adopt a more physically active lifestyle and stimulate the development of effective EXS programs for older PLWH.

DETAILED DESCRIPTION:
Management of older persons living with HIV (PLWH) (≥ 40 years old) is becoming increasingly more complex as a majority is greater than 40 years old. Attempts to improve the quality of life of older PLWH using adjunctive therapeutics to combination antiretroviral therapy (cART) have largely been unsuccessful.

While the impact of physical activity on brain health (assessed by neuropsychological performance and neuroimaging) has been well studied in older healthy HIV uninfected (HIV-) individuals and neurodegenerative conditions, few studies have concentrated on older PLWH. Both clinically and pathophysiologically, HIV associated neurocognitive disorders (HAND) differs from other neurodegenerative disorders seen with aging (e.g. Alzheimer's disease (AD). A positive association relationship between exercise and cognition has been observed in PLWH, but physical activity has been primarily examined using self-report questionnaires that are subjective and not quantitative. To date, no study has focused on the direct effects of exercise on neuropsychological performance or neuroimaging in PLWH.

The objective of this proposal is to conduct a prospective controlled intervention trial to determine if an increase in physical activity through a monitored aerobic and resistance exercise (EXS) program improves brain health in older PLWH. We will quantify physical function (physical activity using cardiorespiratory capacity and actigraphy) and brain function [neuropsychological performance testing and neuroimaging (cerebral blood flow (CBF) and brain volume)] in older physically inactive PLWH at baseline and 26 weeks after randomization to either an EXS or a social-interaction stretching (SIS) program. In addition, we will obtain stool samples, serum markers of neurogenesis, glucose regulation, and systemic inflammation.

A direct impact of these expected outcomes will be the adoption of a more physically active lifestyle by older PLWH and improved EXS guidelines and programs for older PLWH.

ELIGIBILITY:
Inclusion Criteria:

1. age > 40 years old
2. documented history of HIV infection
3. on stable combination antiretroviral therapy (cART) for approximately 3 months with undetectable plasma HIV RNA
4. physically inactive-sedentary lifestyle (approximately <2 hours of exercise/week) and not engaged in regular exercise for approximately 3 months prior to enrollment
5. approximately 9 years of education
6. able to have an MRI
7. able to provide written informed consent (does not have LAR, POA, etc.)

Exclusion Criteria:

1. approximately >2x/week of moderate (or greater) exercise
2. cardiovascular/cerebrovascular disease or pulmonary disease that precludes ability to safely exercise
3. significant neurological disorders (e.g. stroke, head injury with loss of consciousness for >30 minutes, developmental learning disability
4. presence of dementia or behavioral disorders that would prevent ability to follow the protocol
5. alcohol or substance abuse/ dependence within the last 6 months (DSM-4 TR)
6. contraindications to MRI scanning (e.g. claustrophobia, pacemaker)
7. pregnant or breast-feeding
8. unable to provide written informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beau M Ances, MD,PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared when the study has closed.

REFERENCES:
- [Background] Spudich S. HIV and neurocognitive dysfunction. Curr HIV/AIDS Rep. 2013 Sep;10(3):235-43. doi: 10.1007/s11904-013-0171-y. PMID 23860944
- [Background] Spudich S, Gonzalez-Scarano F. HIV-1-related central nervous system disease: current issues in pathogenesis, diagnosis, and treatment. Cold Spring Harb Perspect Med. 2012 Jun;2(6):a007120. doi: 10.1101/cshperspect.a007120. PMID 22675662
- [Background] Clifford DB, Ances BM. HIV-associated neurocognitive disorder. Lancet Infect Dis. 2013 Nov;13(11):976-86. doi: 10.1016/S1473-3099(13)70269-X. PMID 24156898
- [Background] Shah S, Mildvan D. HIV and aging. Curr Infect Dis Rep. 2006 May;8(3):241-7. doi: 10.1007/s11908-006-0065-x. PMID 16643776
- [Background] Valcour V, Paul R. HIV infection and dementia in older adults. Clin Infect Dis. 2006 May 15;42(10):1449-54. doi: 10.1086/503565. Epub 2006 Apr 13. PMID 16619159
- [Background] Hall HI, Song R, Rhodes P, Prejean J, An Q, Lee LM, Karon J, Brookmeyer R, Kaplan EH, McKenna MT, Janssen RS; HIV Incidence Surveillance Group. Estimation of HIV incidence in the United States. JAMA. 2008 Aug 6;300(5):520-9. doi: 10.1001/jama.300.5.520. PMID 18677024
- [Background] Ortega M, Ances BM. Role of HIV in amyloid metabolism. J Neuroimmune Pharmacol. 2014 Sep;9(4):483-91. doi: 10.1007/s11481-014-9546-0. Epub 2014 May 10. PMID 24816714
- [Background] Xu J, Ikezu T. The comorbidity of HIV-associated neurocognitive disorders and Alzheimer's disease: a foreseeable medical challenge in post-HAART era. J Neuroimmune Pharmacol. 2009 Jun;4(2):200-12. doi: 10.1007/s11481-008-9136-0. Epub 2008 Nov 19. PMID 19016329
- [Background] Cohen RA, Seider TR, Navia B. HIV effects on age-associated neurocognitive dysfunction: premature cognitive aging or neurodegenerative disease? Alzheimers Res Ther. 2015 Apr 6;7(1):37. doi: 10.1186/s13195-015-0123-4. eCollection 2015. PMID 25848401
- [Background] Desquilbet L, Jacobson LP, Fried LP, Phair JP, Jamieson BD, Holloway M, Margolick JB. A frailty-related phenotype before HAART initiation as an independent risk factor for AIDS or death after HAART among HIV-infected men. J Gerontol A Biol Sci Med Sci. 2011 Sep;66(9):1030-8. doi: 10.1093/gerona/glr097. Epub 2011 Jun 30. PMID 21719610
- [Background] Justice AC. HIV and aging: time for a new paradigm. Curr HIV/AIDS Rep. 2010 May;7(2):69-76. doi: 10.1007/s11904-010-0041-9. PMID 20425560
- [Background] Justice AC, McGinnis KA, Skanderson M, Chang CC, Gibert CL, Goetz MB, Rimland D, Rodriguez-Barradas MC, Oursler KK, Brown ST, Braithwaite RS, May M, Covinsky KE, Roberts MS, Fultz SL, Bryant KJ; VACS Project Team. Towards a combined prognostic index for survival in HIV infection: the role of 'non-HIV' biomarkers. HIV Med. 2010 Feb;11(2):143-51. doi: 10.1111/j.1468-1293.2009.00757.x. Epub 2009 Sep 14. PMID 19751364
- [Background] Onen NF, Agbebi A, Shacham E, Stamm KE, Onen AR, Overton ET. Frailty among HIV-infected persons in an urban outpatient care setting. J Infect. 2009 Nov;59(5):346-52. doi: 10.1016/j.jinf.2009.08.008. Epub 2009 Aug 23. PMID 19706308
- [Background] Casau NC. Perspective on HIV infection and aging: emerging research on the horizon. Clin Infect Dis. 2005 Sep 15;41(6):855-63. doi: 10.1086/432797. Epub 2005 Jul 28. PMID 16107986
- [Background] Ngandu T, Lehtisalo J, Solomon A, Levalahti E, Ahtiluoto S, Antikainen R, Backman L, Hanninen T, Jula A, Laatikainen T, Lindstrom J, Mangialasche F, Paajanen T, Pajala S, Peltonen M, Rauramaa R, Stigsdotter-Neely A, Strandberg T, Tuomilehto J, Soininen H, Kivipelto M. A 2 year multidomain intervention of diet, exercise, cognitive training, and vascular risk monitoring versus control to prevent cognitive decline in at-risk elderly people (FINGER): a randomised controlled trial. Lancet. 2015 Jun 6;385(9984):2255-63. doi: 10.1016/S0140-6736(15)60461-5. Epub 2015 Mar 12. PMID 25771249
- [Background] Baker LD, Frank LL, Foster-Schubert K, Green PS, Wilkinson CW, McTiernan A, Cholerton BA, Plymate SR, Fishel MA, Watson GS, Duncan GE, Mehta PD, Craft S. Aerobic exercise improves cognition for older adults with glucose intolerance, a risk factor for Alzheimer's disease. J Alzheimers Dis. 2010;22(2):569-79. doi: 10.3233/JAD-2010-100768. PMID 20847403
- [Background] Damirchi A, Tehrani BS, Alamdari KA, Babaei P. Influence of aerobic training and detraining on serum BDNF, insulin resistance, and metabolic risk factors in middle-aged men diagnosed with metabolic syndrome. Clin J Sport Med. 2014 Nov;24(6):513-8. doi: 10.1097/JSM.0000000000000082. PMID 24662570
- [Background] Balsamo S, Willardson JM, Frederico Sde S, Prestes J, Balsamo DC, Dahan da CN, Dos Santos-Neto L, Nobrega OT. Effectiveness of exercise on cognitive impairment and Alzheimer's disease. Int J Gen Med. 2013 May 24;6:387-91. doi: 10.2147/IJGM.S35315. Print 2013. PMID 23737675
- [Background] Rao AK, Chou A, Bursley B, Smulofsky J, Jezequel J. Systematic review of the effects of exercise on activities of daily living in people with Alzheimer's disease. Am J Occup Ther. 2014 Jan-Feb;68(1):50-6. doi: 10.5014/ajot.2014.009035. PMID 24367955
- [Background] Walker JM, Klakotskaia D, Ajit D, Weisman GA, Wood WG, Sun GY, Serfozo P, Simonyi A, Schachtman TR. Beneficial effects of dietary EGCG and voluntary exercise on behavior in an Alzheimer's disease mouse model. J Alzheimers Dis. 2015;44(2):561-72. doi: 10.3233/JAD-140981. PMID 25318545
- [Background] Dufour CA, Marquine MJ, Fazeli PL, Henry BL, Ellis RJ, Grant I, Moore DJ; HNRP Group. Physical exercise is associated with less neurocognitive impairment among HIV-infected adults. J Neurovirol. 2013 Oct;19(5):410-7. doi: 10.1007/s13365-013-0184-8. Epub 2013 Aug 10. PMID 23934585
- [Background] Fazeli PL, Woods SP, Heaton RK, Umlauf A, Gouaux B, Rosario D, Moore RC, Grant I, Moore DJ; HNRP Group. An active lifestyle is associated with better neurocognitive functioning in adults living with HIV infection. J Neurovirol. 2014 Jun;20(3):233-42. doi: 10.1007/s13365-014-0240-z. Epub 2014 Feb 20. PMID 24554483
- [Background] Fillipas S, Oldmeadow LB, Bailey MJ, Cherry CL. A six-month, supervised, aerobic and resistance exercise program improves self-efficacy in people with human immunodeficiency virus: a randomised controlled trial. Aust J Physiother. 2006;52(3):185-90. doi: 10.1016/s0004-9514(06)70027-7. PMID 16942453
- [Background] Mapstone M, Hilton TN, Yang H, Guido JJ, Luque AE, Hall WJ, Dewhurst S, Shah K. Poor Aerobic Fitness May Contribute to Cognitive Decline in HIV-infected Older Adults. Aging Dis. 2013 Aug 27;4(6):311-9. doi: 10.14336/AD.2013.0400311. eCollection 2013. PMID 24307964
- [Background] Mattson MP. Exercise and the brain: a slap on the HAND. J Neurovirol. 2013 Oct;19(5):407-9. doi: 10.1007/s13365-013-0208-4. Epub 2013 Sep 27. No abstract available. PMID 24072548
- [Background] Rodrigues AM, O'Brien N, French DP, Glidewell L, Sniehotta FF. The question-behavior effect: genuine effect or spurious phenomenon? A systematic review of randomized controlled trials with meta-analyses. Health Psychol. 2015 Jan;34(1):61-78. doi: 10.1037/hea0000104. Epub 2014 Aug 18. PMID 25133835
- [Background] Gill AJ, Kolson DL. Chronic inflammation and the role for cofactors (hepatitis C, drug abuse, antiretroviral drug toxicity, aging) in HAND persistence. Curr HIV/AIDS Rep. 2014 Sep;11(3):325-35. doi: 10.1007/s11904-014-0210-3. PMID 24929842
- [Background] Rosenfield PL. The potential of transdisciplinary research for sustaining and extending linkages between the health and social sciences. Soc Sci Med. 1992 Dec;35(11):1343-57. doi: 10.1016/0277-9536(92)90038-r. PMID 1462174
- [Background] Thorpe KE, Zwarenstein M, Oxman AD, Treweek S, Furberg CD, Altman DG, Tunis S, Bergel E, Harvey I, Magid DJ, Chalkidou K. A pragmatic-explanatory continuum indicator summary (PRECIS): a tool to help trial designers. CMAJ. 2009 May 12;180(10):E47-57. doi: 10.1503/cmaj.090523. Epub 2009 Apr 16. No abstract available. PMID 19372436
- [Background] Masters MC, Ances BM. Role of neuroimaging in HIV-associated neurocognitive disorders. Semin Neurol. 2014 Feb;34(1):89-102. doi: 10.1055/s-0034-1372346. Epub 2014 Apr 8. PMID 24715492
- [Derived] Cooley SA, Ferreiro A, Nelson B, Sukhum K, Westerhaus E, Petersen K, Fox JR, Rosenow A, Sorensen C, Vaida F, Reeds DN, Tarr PI, Dantas G, Ances BM. A randomized controlled trial to unveil the influence of an exercise intervention on brain integrity and gut microbiome structure in individuals with HIV. AIDS. 2026 Jan 1;40(1):24-34. doi: 10.1097/QAD.0000000000004346. Epub 2025 Sep 17. PMID 40965137
- [Derived] Cooley S, Nelson BM, Rosenow A, Westerhaus E, Cade WT, Reeds DN, Vaida F, Yarasheski KE, Paul RH, Ances BM. Exercise Training to Improve Brain Health in Older People Living With HIV: Study Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Mar 21;12:e41421. doi: 10.2196/41421. PMID 36943345

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from local clinics as well as a participant registry. Recruitment started in July of 2015 and concluded in November of 2020. There was a pause in recruitment due to the COVID-19 Pandemic from March 2020 through August 2020, and then was terminated early due to a rise in cases in our area in November 2020. A total of 462 were initially screened for the study & 75 were initially enrolled in the study. Out of those 75, a total of 65 were randomized into the intervention.
Groups:
- Exercise (EXS): All EXS sessions will be held at the WUSTL medical campus. Sessions will be offered weekdays. Each session will start with range of motion exercises. Participants will follow an individualized exercise training prescription based on baseline cardiovascular testing. Individual aerobic exercise intensity is based on % of maximum HR achieved during the baseline cardiorespiratory fitness test. The target EXS HR will start at 50% and progress to 85% HR reserve. During aerobic EXS, a battery-operated HR monitor will monitor HR. Exercise intensity & duration will be increased as the participant acclimates to the exercise prescription. Adaptation is determined when a given exercise intensity yields a lower HR than prior sessions conducted at the same intensity.
  The resistance EXS training component will follow aerobic EXS & will consist of 4 upper & 3 lower body routines. A combination of guided-motion machines & free weights will be used. Voluntary maximum strength will be measured during the first 4 sessions on each station. The program will initially consist of 1-2 sets of each exercise while lifting a weight that causes muscle fatigue after 8-10 repetitions. The trainer will monitor each participant's exercise response & when the participant can comfortably lift the weight for 12 repetitions on any exercise, the weight will be increased to cause the muscle group to fatigue after 8 repetitions. This progressive 8-12 repetition cycle is repeated for each exercise over 26 weeks.
Period: Overall Study
Arm/Group | Exercise (EXS) | Social Interaction Stretching (SIS)
Started | 45 | 20
Completed | 33 | 14
Not Completed | 12 | 6

BASELINE CHARACTERISTICS:
Groups:
- Exercise (EXS): EXS sessions will be at an exercise facility at the WUSTL medical campus. Sessions will be offered weekdays. Sessions will start with range of motion EXS. Participants will follow an individualized EXS training prescription based on baseline cardio testing. Individual aerobic EXS intensity is based on % of maximum HR achieved during the baseline cardiorespiratory fitness test. The target EXS HR will start at 50% and progress to 85% HR reserve. During aerobic EXS, HR will be monitored by a battery-operated monitor. EXS intensity & duration will be increased as the participant acclimates to the EXS prescription. Adaptation is determined when a given EXS intensity yields a lower HR than prior sessions conducted at the same intensity.
  Exercise: The resistance EXS training component will follow aerobic exercise and will consist of 4 upper and 3 lower body routines. A combination of guided-motion machines & free weights will be used. Voluntary maximum strength will be measured during the first 4 sessions on each exercise station. The program will initially consist of 1-2 sets of each exercise while lifting a weight that causes muscle fatigue after 8-10 repetitions. The trainer will monitor each participant's EXS response, & when the participant can comfortably lift the weight for 12 repetitions on any exercise, the weight will be increased to cause the muscle group to fatigue after 8 repetitions. This progressive 8-12 repetition cycle is repeated for each exercise over 26 weeks.
- Total: Total of all reporting groups
Arm/Group | Exercise (EXS) | Social Interaction Stretching (SIS) | Total
Number analyzed (Participants) | 45 | 20 | 65
Age, Continuous [Mean (Full Range); unit: years] | 56.5 [41 to 70] | 56.5 [50 to 71] | 56.5 [41 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 2 | 15
  Male | 32 | 18 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 14 | 43
  White | 16 | 6 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 45 | 20 | 65
Education [Mean (Standard Deviation); unit: years] | 12.9 (2.4) | 13.9 (2.2) | 13.2 (2.4)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30.5 (7.0) | 28.9 (5.7) | 29.7 (6.6)
Viral Load Undetectable (<50 copies/mL) [Count of Participants; unit: Participants] — An undetectable viral load is currently recognized as HIV-1 RNA viral load <50 copies/mL. This means there are less than 50 copies of the virus present in a blood sample. This measure is stating how many participants were currently undetectable at the time of enrollment into the study.
  Participants | 45 | 20 | 65
Median recent CD4 T-cell count (cells/mm3) (IQR) [Median (Inter-Quartile Range); unit: cells/mm3] — CD4 T cells are a type of lymphocyte. CD4 T lymphocytes (CD4 cells) help coordinate the immune response by stimulating other immune cells, such as macrophages, B lymphocytes (B cells), and CD8 T lymphocytes (CD8 cells), to fight infection. HIV weakens the immune system by destroying CD4 cells.
  The median recent CD4 T-Cell count is the value separating the higher half from the lower half of a data sample.
  cells/mm3 | 581 [474 to 817] | 561 [362 to 771] | 578 [450 to 789]
Median CD4 nadir T-cell count (cells/mm3) (IQR) [Median (Inter-Quartile Range); unit: cells/mm3] — CD4 Nadir refers to the lowest historical value for CD4 T cell count. Research has shown that a Nadir CD4 T-cell count is a predictor of negative outcomes in HIV -infected patients.
  The median CD4 Nadir is the value separating the higher half from the lower half the data sample.
  cells/mm3 | 195 [22 to 312] | 47 [25 to 358] | 179.5 [24 to 300]
Median CD8 T-cell count (cells/mm3) (IQR) [Median (Inter-Quartile Range); unit: cells/mm3] — CD8 T cells are an indication of active HIV infection. The lower the CD8 the less active virus is in the system. The median is the value separating the higher half from the lower half of a data sample.
  cells/mm3 | 809 [489 to 1079] | 689 [577 to 1035] | 785 [520 to 1085]
Mean duration of HIV infection (in months) (SD) [Mean (Standard Deviation); unit: Months of Infection] | 225.4 (117.6) | 259.0 (94.3) | 235.4 (109.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Cognition From Baseline to Follow up, in Exercise Group vs. Stretching Group
Description: This measure examines the global z-score which is an average of all the individual cognitive test z scores. We looked at changes in global Z-scores from baseline to follow-up (6 months). A Z-score of 0 represents the population mean. Z-scores are considered to be better when they are above the mean and represent a better outcome.
Time Frame: 6 months
Population: All participants who completed cognitive testing at baseline and 6 months.
Measure: Mean (Standard Deviation); unit: z-score
Groups:
- Exercise (EXS): All Exercise sessions will be at an exercise facility at the WUSTL medical campus. Sessions will be offered weekdays. Sessions will start with range of motion exercises. Participants will follow an individualized EXS training prescription based on baseline cardio testing. Individual aerobic EXS intensity is based on % of maximum HR achieved during the baseline cardiorespiratory fitness test. The target EXS HR will start at 50% and progress to 85% HR reserve. During aerobic EXS, HR will be monitored by a battery-operated HR monitor. EXS intensity & duration will be increased as the participant acclimates to the EXS prescription. Adaptation is determined when a given EXS intensity yields a lower HR than prior sessions conducted at the same intensity.
  Exercise: The resistance EXS training component will follow aerobic EXS & will consist of 4 upper and 3 lower body routines. A combination of guided-motion machines and free weights will be used. Voluntary maximum strength will be measured during the first 4 sessions on each EXS station. The program will initially consist of 1-2 sets of each EXS while lifting a weight that causes muscle fatigue after 8-10 repetitions. The trainer will monitor each participant's EXS response, and when the participant can comfortably lift the weight for 12 repetitions on any EXS, the weight will be increased to cause the muscle group to fatigue after 8 repetitions. This progressive 8-12 repetition cycle is repeated for each EXS over 26 weeks.
- Social Interaction Stretching (SIS): This group will serve as a control group against which to gauge the effects of aerobic and resistance training on cognitive function. Participants in this group will follow the same schedule and format as the Exercise group. These participants will be supervised by the same trainer and will receive the same amount of attention and class interaction as participants in the Exercise program. These Stretching participants will receive instructions on stretching, range of motion, limbering, and toning; but the intensity will be far less than that achieved in the Exercise classes. Activities will focus on flexibility enhancement. As the participant's level of flexibility increases, stretches with increasing levels of difficulty will be incorporated into the program.
  Stretching and Social Interaction: Participants will receive instructions on stretching, range of motion, limbering, and toning. Activities will focus on flexibility enhancement. Along with the stretching and flexibility, this group will have a social interaction component. They will have discussions and interact with trainers and coordinators during all their sessions. These participants will be supervised by the same trainer and will receive the same amount of attention and class interaction as participants in the Exercise program.
Arm/Group | Exercise (EXS) | Social Interaction Stretching (SIS)
Number analyzed (Participants) | 33 | 14
z-score | .10 (.29) | .20 (.33)
Statistical Analysis 1: Comparison: Exercise (EXS) vs Social Interaction Stretching (SIS); Test type: Superiority; p = 0.31, ANOVA; Mean Difference (Net) = 0.15, 95% CI 2-sided [.05 to .25]

2. Primary Outcome: Changes in Brain Structural/Functional Measures in Older PLWH
Description: The Investigators will assess if an EXS program improves brain structure and function more than a SIS program in older sedentary PLWH. Changes in brain volumetrics (total cortex volume) at baseline (BL) and 26 weeks will be compared between EXS and SIS groups.
Time Frame: 26 weeks
Population: Participants from both the Exercise and Stretching group's MRIs were analyzed for cortical volume change from pre-intervention to post-intervention.
Measure: Mean (Standard Deviation); unit: mm^3
Groups:
- Exercise (EXS): All EXS sessions will be at an exercise facility at the WUSTL medical campus. Sessions will be offered weekdays. Sessions will start with range of motion EXS. Participants will follow an individualized EXS training prescription based on baseline cardio testing. Individual aerobic EXS intensity is based on % of maximum HR achieved during the baseline cardiorespiratory fitness test. The target EXS HR will start at 50% and progress to 85% HR reserve. During aerobic EXS, a battery-operated HR monitor will monitor HR. EXS intensity & duration will be increased as the participant acclimates to the EXS prescription. Adaptation is determined when a given EXS intensity yields a lower HR than prior sessions conducted at the same intensity.
  Exercise: The resistance EXS training component will follow aerobic EXS and will consist of 4 upper and 3 lower body routines. A combination of guided-motion machines and free weights will be used. Voluntary maximum strength will be measured during the first 4 sessions on each exercise station. The program will initially consist of 1-2 sets of each EXS while lifting a weight that causes muscle fatigue after 8-10 repetitions. The trainer will monitor each participant's EXS response, and when the participant can comfortably lift the weight for 12 repetitions on any EXS, the weight will be increased to cause the muscle group to fatigue after 8 repetitions. This progressive 8-12 repetition cycle is repeated for each EXS over 26 weeks.
Arm/Group | Exercise (EXS) | Social Interaction Stretching (SIS)
Number analyzed (Participants) | 33 | 14
mm^3 | -546.1 (10358) | 366.6 (8102)
Statistical Analysis 1: Comparison: Exercise (EXS) vs Social Interaction Stretching (SIS); Change in Global CBF in EXS vs. SIS; Test type: Superiority; p = .24, ANOVA; Mean Difference (Net) = 1.42
Statistical Analysis 2: Comparison: Exercise (EXS); Change in Strength & Change in Frontal Brain Volume in EXS; Test type: Other; p = .02, Regression, Linear; Slope = 0.41
Statistical Analysis 3: Comparison: Exercise (EXS); Changes in Brain Volumes associated with changes Memory Performance in EXS; Test type: Other; p = 0.02, Regression, Linear; Slope = 0.40

3. Primary Outcome: Change in Level of Daily Activity
Description: Investigators will examine the amount of change in daily activity based on 7-day actigraphy at baseline and then again at follow-up (26 weeks later). Daily activity is measured using an actigraph that participants wear on their wrist and it measures the amount of time spent in sedentary, slightly active, moderately active, vigorously active or very vigorously active categories.
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: Average Minutes per Day
Arm/Group | Exercise (EXS) | Social Interaction Stretching (SIS)
Number analyzed (Participants) | 33 | 14
Average Minutes per Day | -23.9 (114.8) | -5.3 (98.9)
Statistical Analysis 1: Comparison: Exercise (EXS); Increases in Time Spent in MVPA and Increased Learning Performance in EXS; Test type: Other; p = .005, Regression, Linear; Slope = .47

ADVERSE EVENTS:
Time Frame: Through study completion, an average of approximately 6 months per participant.
Description: Adverse events were defined by the clinicaltrials.gov definitions.
Groups:
- Exercise (EXS): All EXS sessions will be at a facility at the WUSTL medical campus. Sessions will be offered weekdays. Each session will start with range of motion EXS. Participants will follow an individualized EXS training prescription based on baseline cardiovascular testing. Individual aerobic EXS intensity is based on % of maximum HR achieved during the baseline cardiorespiratory fitness test. The target EXS HR will start at 50% and progress to 85% HR reserve. During aerobic exercise, a battery-operated HR monitor will monitor HR. Exercise intensity & duration will be increased as the participant acclimates to the EXS prescription. Adaptation is determined when a given EXS intensity yields a lower HR than prior sessions conducted at the same intensity.
  Exercise: The resistance EXS training component will follow aerobic EXS and will consist of 4 upper and 3 lower body routines. A combination of guided-motion machines and free weights will be used. Voluntary maximum strength will be measured during the first 4 sessions on each EXS station. The program will initially consist of 1-2 sets of each exercise while lifting a weight that causes muscle fatigue after 8-10 repetitions. The trainer will monitor each participant's EXS response, and when the participant can comfortably lift the weight for 12 repetitions on any EXS, the weight will be increased to cause the muscle group to fatigue after 8 repetitions. This progressive 8-12 repetition cycle is repeated for each EXS over 26 weeks.
Arm/Group | Exercise (EXS) | Social Interaction Stretching (SIS)
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/20
Other Adverse Events (participants affected / at risk) | 0/45 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/34/NCT02663934/Prot_SAP_002.pdf
  • Informed Consent Form (2020-07-23): https://cdn.clinicaltrials.gov/large-docs/34/NCT02663934/ICF_001.pdf